CLINICAL TRIAL: NCT01110499
Title: Safety and Efficacy of AGN-210961 Ophthalmic Solution Compared With Bimatoprost Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 210961-002
Record Dates: First submitted 2010-04-23; First posted 2010-04-26 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-07

CONDITIONS: Ocular Hypertension; Primary Open-Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part 1, AGN-210961 Formulation 1 (Experimental): AGN-210961 Formulation 1 in one eye and bimatoprost ophthalmic solution 0.03% in the other eye once daily for 7 days.
  Interventions: Drug: AGN-210961 Formulation 1
- Part 1, AGN-210961 Formulation 2 (Experimental): AGN-210961 Formulation 2 in one eye and bimatoprost ophthalmic solution 0.03% in the other eye once daily for 7 days.
  Interventions: Drug: AGN-210961 Formulation 2
- Part 1, AGN-210961 Formulation 3 (Experimental): AGN-210961 Formulation 3 in one eye and bimatoprost ophthalmic solution 0.03% in the other eye once daily for 7 days.
  Interventions: Drug: AGN-210961 Formulation 3
- Part 1, AGN-210961 Formulation 4 (Experimental): AGN-210961 Formulation 4 in one eye and bimatoprost ophthalmic solution 0.03% in the other eye once daily for 7 days.
  Interventions: Drug: AGN-210961 Formulation 4
- Part 1, AGN-210961 Formulation 5 (Experimental): AGN-210961 Formulation 5 in one eye and bimatoprost ophthalmic solution 0.03% in the other eye once daily for 7 days.
  Interventions: Drug: AGN-210961 Formulation 5
- Part 1, AGN-210961 Formulation 6 (Experimental): AGN-210961 Formulation 6 in one eye and bimatoprost ophthalmic solution 0.03% in the other eye once daily for 7 days.
  Interventions: Drug: AGN-210961 Formulation 6
- Part 2, AGN-210961 Formulation 7 (Experimental): AGN-210961 Formulation 7 in both eyes once daily for 4 weeks.
  Interventions: Drug: AGN-210961 Formulation 7
- Part 2, bimatoprost ophthalmic solution 0.03% (Active Comparator): bimatoprost ophthalmic solution 0.03% in both eyes once daily for 4 weeks.
  Interventions: Drug: bimatoprost ophthalmic solution 0.03%

INTERVENTIONS:
Drug: AGN-210961 Formulation 1 — AGN-210961 Formulation 1 in one eye once daily for 7 days.
  Arms: Part 1, AGN-210961 Formulation 1
Drug: AGN-210961 Formulation 2 — AGN-210961 Formulation 2 in one eye once daily for 7 days.
  Arms: Part 1, AGN-210961 Formulation 2
Drug: AGN-210961 Formulation 3 — AGN-210961 Formulation 3 in one eye once daily for 7 days.
  Arms: Part 1, AGN-210961 Formulation 3
Drug: AGN-210961 Formulation 4 — AGN-210961 Formulation 4 in one eye once daily for 7 days.
  Arms: Part 1, AGN-210961 Formulation 4
Drug: AGN-210961 Formulation 5 — AGN-210961 Formulation 5 in one eye once daily for 7 days.
  Arms: Part 1, AGN-210961 Formulation 5
Drug: AGN-210961 Formulation 6 — AGN-210961 Formulation 6 in one eye once daily for 7 days.
  Arms: Part 1, AGN-210961 Formulation 6
Drug: AGN-210961 Formulation 7 — AGN-210961 Formulation 7 in both eyes once daily for 4 weeks.
  Arms: Part 2, AGN-210961 Formulation 7
Drug: bimatoprost ophthalmic solution 0.03% — bimatoprost ophthalmic solution 0.03% (LUMIGAN®) in both eyes once daily for 4 weeks.
  Other Names: LUMIGAN®
  Arms: Part 2, bimatoprost ophthalmic solution 0.03%

SUMMARY:
This study has 2 parts. Part 1 will evaluate the safety and IOP effects of 6 formulations of AGN-210961 ophthalmic solution in the study eye and bimatoprost ophthalmic solution 0.03% in the fellow eye for 7 consecutive days. Part 2 will evaluate the safety and IOP effects of a formulation (to be selected from part 1) of AGN-210961 in both eyes compared to bimatoprost ophthalmic solution 0.03% for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Ocular hypertension or primary open-angle glaucoma in each eye

Exclusion Criteria:

* Any active ocular disease
* Anticipated wearing of contact lenses during study
* Anticipated use of artificial tears during study
* Contraindication to pupil dilatation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-part study. Patients were enrolled in and completed Part 1 of the study. Then, based on a review of the data from Part 1, a different formulation was selected for Part 2 (Formulation 7). New patients were then enrolled in Part 2 of the study. No patients from Part 1 were enrolled in Part 2 of the study.
Groups:
- Part 2, AGN-210961 Formulation 7: AGN-210961 Formulation 7 (a different formulation from those used in Part 1) in both eyes once daily for 4 weeks.
Period: Overall Study
Arm/Group | Part 1, AGN-210961 Formulation 1 | Part 1, AGN-210961 Formulation 2 | Part 1, AGN-210961 Formulation 3 | Part 1, AGN-210961 Formulation 4 | Part 1, AGN-210961 Formulation 5 | Part 1, AGN-210961 Formulation 6 | Part 2, AGN-210961 Formulation 7 | Part 2, Bimatoprost Ophthalmic Solution 0.03%
Started | 14 | 14 | 14 | 14 | 14 | 14 | 39 | 40
Completed | 14 | 14 | 14 | 14 | 14 | 14 | 39 | 40
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, AGN-210961 Formulation 1 | Part 1, AGN-210961 Formulation 2 | Part 1, AGN-210961 Formulation 3 | Part 1, AGN-210961 Formulation 4 | Part 1, AGN-210961 Formulation 5 | Part 1, AGN-210961 Formulation 6 | Part 2, AGN-210961 Formulation 7 | Part 2, Bimatoprost Ophthalmic Solution 0.03% | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 39 | 40 | 163
Age, Customized [Number; unit: Participants]
  <45 years | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 4
  45 to 65 years | 11 | 3 | 6 | 8 | 6 | 7 | 18 | 23 | 82
  >65 years | 3 | 10 | 7 | 5 | 8 | 7 | 21 | 16 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 10 | 9 | 7 | 7 | 24 | 27 | 105
  Male | 2 | 5 | 4 | 5 | 7 | 7 | 15 | 13 | 58

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. Data are recorded at Hours 0, 2, 4, 6, 8, and 12. A negative number change from Baseline indicated a reduction in IOP (improvement). Data for bimatoprost-treated eyes are combined across groups.
Time Frame: Baseline, Day 7
Population: Safety Population: all treated patients
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Units Other Than Participants: Eyes
Groups:
- Part 1, AGN-210961 Formulation 1: AGN-210961 Formulation 1 in one eye once daily for 7 days.
- Part 1, AGN-210961 Formulation 2: AGN-210961 Formulation 2 in one eye once daily for 7 days.
- Part 1, AGN-210961 Formulation 3: AGN-210961 Formulation 3 in one eye once daily for 7 days.
- Part 1, AGN-210961 Formulation 4: AGN-210961 Formulation 4 in one eye once daily for 7 days.
- Part 1, AGN-210961 Formulation 5: AGN-210961 Formulation 5 in one eye once daily for 7 days.
- Part 1, AGN-210961 Formulation 6: AGN-210961 Formulation 6 in one eye once daily for 7 days.
- Part 1, Bimatoprost Ophthalmic Solution 0.03%: bimatoprost ophthalmic solution 0.03% in the other eye in all Part 1 treatment groups once daily for 7 days.
Arm/Group | Part 1, AGN-210961 Formulation 1 | Part 1, AGN-210961 Formulation 2 | Part 1, AGN-210961 Formulation 3 | Part 1, AGN-210961 Formulation 4 | Part 1, AGN-210961 Formulation 5 | Part 1, AGN-210961 Formulation 6 | Part 1, Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 84
Number analyzed (Eyes) | 14 | 14 | 14 | 14 | 14 | 14 | 84
Millimeters of Mercury (mmHg)
  Baseline - Hour 0 | 25.4 (2.5) | 25.6 (2.71) | 24.3 (1.94) | 26.7 (3.60) | 24.4 (1.54) | 25.3 (2.23) | 25.3 (2.82)
  Baseline - Hour 2 | 23.1 (2.18) | 23.5 (2.53) | 23.6 (2.64) | 23.6 (3.27) | 23.1 (3.49) | 24.1 (3.25) | 23.4 (2.83)
  Baseline - Hour 4 | 23.5 (2.53) | 23.1 (2.55) | 23.6 (3.64) | 23.0 (3.72) | 23.1 (2.46) | 23.7 (2.49) | 23.2 (2.76)
  Baseline - Hour 6 | 22.0 (2.53) | 22.0 (2.46) | 24.4 (4.43) | 21.9 (3.88) | 22.1 (2.60) | 22.4 (2.72) | 22.5 (3.33)
  Baseline - Hour 8 | 21.6 (2.84) | 21.3 (2.58) | 23.2 (3.87) | 22.1 (4.04) | 22.2 (2.83) | 22.9 (2.95) | 22.3 (3.18)
  Baseline - Hour 12 | 22.1 (2.98) | 21.6 (3.03) | 21.8 (3.86) | 21.6 (4.24) | 21.3 (1.98) | 20.8 (2.44) | 21.5 (3.10)
  Change from Baseline at Day 7- Hour 0 | -6.1 (4.22) | -6.3 (4.24) | -5.9 (4.36) | -6.0 (3.87) | -5.2 (3.79) | -5.6 (3.16) | -6.3 (3.66)
  Change from Baseline at Day 7- Hour 2 | -5.3 (3.00) | -6.6 (2.88) | -6.0 (2.72) | -5.6 (2.80) | -5.3 (3.97) | -5.2 (3.71) | -5.0 (3.06)
  Change from Baseline at Day 7- Hour 4 | -6.6 (4.27) | -4.5 (2.45) | -6.3 (4.35) | -4.0 (2.48) | -5.2 (3.60) | -5.2 (3.68) | -5.1 (2.79)
  Change from Baseline at Day 7 - Hour 6 | -5.6 (2.23) | -4.5 (3.03) | -6.7 (4.05) | -3.2 (3.49) | -5.1 (2.23) | -4.7 (2.63) | -5.5 (2.92)
  Change from Baseline at Day 7- Hour 8 | -5.9 (2.91) | -4.8 (2.45) | -5.8 (3.31) | -4.4 (2.49) | -5.5 (3.28) | -4.9 (3.94) | -6.2 (2.99)
  Change from Baseline at Day 7- Hour 12 | -5.4 (3.77) | -4.9 (3.39) | -4.8 (3.69) | -4.8 (3.41) | -3.7 (3.88) | -3.7 (3.21) | -5.6 (2.73)

2. Primary Outcome: Part 2: Change From Baseline in Average Eye Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. Average IOP is the average of the 2 eyes for each patient at each time point. A negative number change from Baseline indicates a reduction in IOP (improvement). Data are recorded at Hours 0, 2, 4, 6, 8, and 12.
Time Frame: Baseline, Day 29
Population: Modified Intent to Treat: all randomized and treated patients who provided IOP data for baseline and at least one postbaseline hour 0 assessment
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Part 2, AGN-210961 Formulation 7 | Part 2, Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 39 | 40
Millimeters of Mercury (mmHg)
  Baseline - Hour 0 | 24.63 (2.526) | 24.62 (2.465)
  Baseline - Hour 2 | 23.40 (2.072) | 23.70 (3.182)
  Baseline - Hour 4 | 22.25 (2.449) | 22.51 (3.507)
  Baseline - Hour 6 | 21.97 (2.264) | 22.38 (3.492)
  Baseline - Hour 8 | 21.28 (2.896) | 21.48 (3.354)
  Baseline - Hour 12 | 20.72 (3.162) | 20.94 (3.549)
  Change from Baseline at Day 29 - Hour 0 | -7.44 (3.173) | -8.63 (3.399)
  Change from Baseline at Day 29 - Hour 2 | -7.40 (3.269) | -8.51 (3.752)
  Change from Baseline at Day 29 - Hour 4 | -6.25 (3.521) | -7.39 (3.993)
  Change from Baseline at Day 29 - Hour 6 | -6.31 (3.625) | -6.92 (3.808)
  Change from Baseline at Day 29 - Hour 8 | -6.15 (3.856) | -6.31 (4.056)
  Change from Baseline at Day 29 - Hour 12 | -5.74 (4.086) | -5.10 (4.054)

ADVERSE EVENTS:
Description: AEs and SAEs are reported for all treated patients. In Part 1, ocular AEs for bimatoprost treated eye are noted in "Part 1, bimatoprost 0.03% treated eye" only and those for AGN-210961 Formulations 1-6 eyes are noted in "Part 1, AGN-210961 Formulations 1-6". In Part 1, non-ocular AEs are reported only in "Part 1, AGN-210961 Formulations 1-6" arms.
Groups:
- Part 1, Bimatoprost Ophthalmic Solution 0.03% Treated Eye: bimatoprost ophthalmic solution 0.03% in the non-study eye once daily for 7 days (all bimatoprost ophthalmic solution 0.03% treated eyes in Part 1 combined).
Arm/Group | Part 1, AGN-210961 Formulation 1 | Part 1, AGN-210961 Formulation 2 | Part 1, AGN-210961 Formulation 3 | Part 1, AGN-210961 Formulation 4 | Part 1, AGN-210961 Formulation 5 | Part 1, AGN-210961 Formulation 6 | Part 1, Bimatoprost Ophthalmic Solution 0.03% Treated Eye | Part 2, AGN-210961 Formulation 7 | Part 2, Bimatoprost Ophthalmic Solution 0.03%
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/84 | 1/39 | 1/40
Other Adverse Events (participants affected / at risk) | 10/14 | 9/14 | 10/14 | 6/14 | 7/14 | 5/14 | 53/84 | 29/39 | 19/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, AGN-210961 Formulation 1 (N=14) | Part 1, AGN-210961 Formulation 2 (N=14) | Part 1, AGN-210961 Formulation 3 (N=14) | Part 1, AGN-210961 Formulation 4 (N=14) | Part 1, AGN-210961 Formulation 5 (N=14) | Part 1, AGN-210961 Formulation 6 (N=14) | Part 1, Bimatoprost Ophthalmic Solution 0.03% Treated Eye (N=84) | Part 2, AGN-210961 Formulation 7 (N=39) | Part 2, Bimatoprost Ophthalmic Solution 0.03% (N=40)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip and/or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, AGN-210961 Formulation 1 (N=14) | Part 1, AGN-210961 Formulation 2 (N=14) | Part 1, AGN-210961 Formulation 3 (N=14) | Part 1, AGN-210961 Formulation 4 (N=14) | Part 1, AGN-210961 Formulation 5 (N=14) | Part 1, AGN-210961 Formulation 6 (N=14) | Part 1, Bimatoprost Ophthalmic Solution 0.03% Treated Eye (N=84) | Part 2, AGN-210961 Formulation 7 (N=39) | Part 2, Bimatoprost Ophthalmic Solution 0.03% (N=40)
Conjunctival Hyperaemia (Eye disorders) | 5 | 5 | 6 | 3 | 3 | 3 | 42 | 16 | 16
Punctate Keratitis (Eye disorders) | 4 | 3 | 5 | 2 | 2 | 0 | 16 | 7 | 5
Corneal thickening (Eye disorders) | 2 | 3 | 3 | 1 | 2 | 2 | 0 | 22 | 1
Photophobia (Eye disorders) | 2 | 1 | 2 | 1 | 2 | 0 | 4 | 11 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 2 | 2 | 0 | 2 | 1 | 2 | 7 | 1
Eye Pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 3
Iritis (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 1
Eye Pruritus (Eye disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 5 | 2 | 5
Bundle Branch Block Right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foreign Body Sensation in Eyes (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 4
Hemicephalalgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.